CLINICAL TRIAL: NCT03206177
Title: Feasibility IB Trial of Paclitaxel/Carboplatin + Galunisertib (a Small Molecule Inhibitor of the Kinase Domain of Type 1 TGF-B Receptor) in Patients With Newly Diagnosed, Persistent or Recurrent Carcinosarcoma of the Uterus or Ovary
Brief Title: Paclitaxel/Carboplatin + Galunisertib for Patients With Carcinosarcoma of the Uterus or Ovary
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-EXIST-001
Record Dates: First submitted 2017-06-01; First posted 2017-07-02 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-03

CONDITIONS: Carcinosarcoma, Ovarian
MeSH Terms: conditions — Carcinosarcoma | interventions — LY-2157299; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Paclitaxel/Carboplatin + Galunisertib (Experimental): Patients will receive the following in every cycle (1 cycle=28days).
  * Paclitaxel - 175 mg/m2 over 3 hours via IV on Day 1
  * Carboplatin - AUC 6* (or AUC 5*) over 1 hour via IV on Day 1
  * Galunisertib - 150mg orally twice a day on Days 4-17
  Interventions: Drug: Galunisertib; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Galunisertib — Galunisertib 150mg po BID day 4-17
Drug: Paclitaxel — IV Day 1: Paclitaxel 175 mg/m2 over 3 hours
Drug: Carboplatin — IV Day 1: Carboplatin AUC 6* over 1 hour (or 5* if prior radiation therapy)

SUMMARY:
This is a Phase 1 B feasibility trial with Galunsertib, a TGFβ inhibitor, in combination with carboplatin/paclitaxel in patients with newly diagnosed, persistent or recurrent carcinosarcoma of the uterus or ovary. The objective of the study is to determine whether this drug combination is safe for this patient population and to see if it is effective in shrinking cancers, keeping them from growing or helping patients live longer.

DETAILED DESCRIPTION:
Patients who consent to this study will receive treatment for four 28 day cycles unless they are unable to continue study treatment due to toxicity or disease progression. Paclitaxel and carboplatin will be given intravenously on day 1 of each cycle and galunisertib in pill form on days 4-17. No medicine will be given on days 17-28 of each cycle. Patients may have the option of continuing treatment with the study drug if they complete the 4 cycles the study requires. Subjects will receive tests and procedures that are part of regular cancer care as well as those required for the purposes of the study. Blood samples will be taken to monitor the level of study drug in the blood. Patients will have the option of allowing blood and tumor samples to be used for future research.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years old with a diagnosis of primary, recurrent or progressive uterine, ovarian, fallopian tube or peritoneal carcinosarcoma, for whom treatment with combination paclitaxel and carboplatin is recommended.
2. Written informed consent/assent prior to any study-specific procedures
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Tissue available for translational study (paraffin block or new biopsy) .
5. Adequate bone marrow, renal, and hepatic function as defined per protocol.
6. No disease-modifying therapy, including investigational treatments, within 28 days prior to initiation of study treatment.
7. Ability to swallow tablets
8. For Women of child-bearing potential:Willingness to use a highly effective method of contraception during the study and for 6 months following the last dose of galunisertib. Negative beta human chorionic gonadotropin pregnancy test documented within 7 days prior to initiation of study drug.
9. Patient must have measurable disease before the treatment

Exclusion Criteria:

1. Planned radiotherapy during or after the study chemotherapy prior to disease progression.
2. Receipt of chemotherapy or radiation within 28 days of study treatment
3. Have had a major surgical procedure or a significant traumatic injury within 28 days prior to study treatment; Minor procedures such as biopsy within 7 days prior to study treatment are allowed.
4. Active infection that would preclude receipt of chemotherapy
5. Moderate or severe cardiovascular disease per protocol
6. Active pregnancy or lactation
7. Second primary malignancy for which treatment during the study period would be recommended if this cancer were not also present.
8. Prior malignancy requiring treatment within the last 3 years
9. Use of another investigational product or device within 4 weeks of study entry or during study participation.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The patient population for this study only applies to females.
Enrollment: 26 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, MD, Principal Investigator — Obstetrics and Gynecology
Locations (1):
- Stephenson Cancer Center, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single site study conducted at the University of Oklahoma Stephenson Cancer Center enrolled 26 participants between August 2017 and March 2021. The first participant was enrolled on August 23, 2017 and the last participant was enrolled on March 29, 2021.
Pre-assignment Details: Of the 26 enrolled participants, 24 met inclusion criteria (2 participants were screen-fails) and were assigned to the study arm to receive treatment. Of the 24 participants that received treatment, 23 participants were evaluable based on the protocol.
Period: Overall Study
Arm/Group | Paclitaxel/Carboplatin + Galunisertib
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Patients who enrolled in study
Groups:
- Paclitaxel/Carboplatin + Galunisertib: Galunisertib: Galunisertib 150mg po BID day 4-17
  Paclitaxel: Paclitaxel 175 mg/m2 over 3 hours
  Carboplatin: IV day 1 Carboplatin AUC 6* over 1 hour (or 5* if prior radiation therapy)
Arm/Group | Paclitaxel/Carboplatin + Galunisertib
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.96 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 24
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: One patient did not receive baseline weight measurement
  kg/m^2
    number analyzed (Participants) | 23
    (all) | 27.08 (8.40)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Completion of 4 Cycles of CT + GB
Description: Completion of 4 cycles of CT + GB- completion of a cycle will be defined as receiving both carboplatin/paclitaxel and taking ≥75% of the doses of GB for the cycle.
Time Frame: 2 years
Population: Evaluable patients will be defined as patients who receive at least four cycles of study treatment.
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | Paclitaxel/Carboplatin + Galunisertib
Number analyzed (Participants) | 23
proportion of patients | 0.7826 [0.5961 to 0.9102]

2. Secondary Outcome: Median Progression Free Survival (Months)
Description: Progression free survival is defined as time from when the patient is registered on the study until RECIST v1.1 documented disease progression as per the protocol or death.
Time Frame: through study completion, an average of 3 years
Population: Patients who received at least four cycles of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel/Carboplatin + Galunisertib
Number analyzed (Participants) | 23
months | 6.55 [5.42 to 10.81]

3. Secondary Outcome: Median Overall Survival (Months)
Description: Overall survival defined as time from study entry to death
Time Frame: through study completion, an average of 3 years
Population: Patients who received at least four cycles of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel/Carboplatin + Galunisertib
Number analyzed (Participants) | 23
months | 18.91 [10.81 to NA] — The curve that represents the upper confidence limit never crosses below 0.5 and therefore an upper bound for the median value cannot be calculated.

4. Secondary Outcome: Objective Response
Description: Proportion of patients who had RECIST documented partial or complete response. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be ≥ 10 mm when measured by CT and MRI; or ≥ 20 mm when measured by conventional techniques, including plain x-ray. Response was documented per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions.
Time Frame: within three years of study entry
Population: Patients who received four cycles of study drugs
Measure: Number (95% Confidence Interval); unit: proportion of patients with CR/PR
Arm/Group | Paclitaxel/Carboplatin + Galunisertib
Number analyzed (Participants) | 21
proportion of patients with CR/PR | 0.33 [0.15 to 0.57]

ADVERSE EVENTS:
Time Frame: Within 4 years of study entry
Arm/Group | Paclitaxel/Carboplatin + Galunisertib
All-Cause Mortality (participants affected / at risk) | 1/24
Serious Adverse Events (participants affected / at risk) | 11/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel/Carboplatin + Galunisertib (N=24)
ARTRIAL FIBRILLATION (Cardiac disorders) | 1
SMALL BOWEL OBSTRUCTION (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
DEATH (General disorders) | 1
FEVER (General disorders) | 1
NEUTROPENIC FEVER (General disorders) | 1
PULMONARY INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
DRUG INDUCED LIVER INJURY (Injury, poisoning and procedural complications) | 1
LEFT LEG FRACTURE (Musculoskeletal and connective tissue disorders) | 1
STROKE (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
CONFUSION (Psychiatric disorders) | 1
VAGINAL BLEEDING (Reproductive system and breast disorders) | 1
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1
THROMBOEMBOLIC EVENT (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel/Carboplatin + Galunisertib (N=24)
ANEMIA (Blood and lymphatic system disorders) | 4
NEUTROPENIA (Blood and lymphatic system disorders) | 10
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 4
GERD (Gastrointestinal disorders) | 2
INTERMITTENT NAUSEA (Gastrointestinal disorders) | 3
NAUSEA (Gastrointestinal disorders) | 9
VOMITING (Gastrointestinal disorders) | 2
FATIGUE (General disorders) | 11
INFUSION REACTION (General disorders) | 2
INFUSION RELATED REACTION (General disorders) | 2
INTERMITTENT FATIGUE (General disorders) | 2
URINARY TRACT INFECTION (Infections and infestations) | 6
FALL (Injury, poisoning and procedural complications) | 3
ANOREXIA (Metabolism and nutrition disorders) | 4
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
DIZZINESS (Nervous system disorders) | 3
DYSGEUSIA (Nervous system disorders) | 3
HEADACHE (Nervous system disorders) | 3
NEUROPATHY (Nervous system disorders) | 13
PERIPHERAL NEUROPATHY (Nervous system disorders) | 2
INSOMNIA (Psychiatric disorders) | 2
VAGINAL BLEEDING (Reproductive system and breast disorders) | 2
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 2
RASH (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT03206177/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT03206177/SAP_001.pdf
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT03206177/ICF_002.pdf